CLINICAL TRIAL: NCT04192552
Title: Perioperative Anticoagulant (Dabigatran, Rivaroxaban, or Apixaban) Use for Elective Surgery/Procedure Evaluation in Patients With Atrial Fibrillation (AF) Part 2 Randomized Control Trial Pilot
Brief Title: Perioperative Anticoagulant Use for Surgery Evaluation Study Part 2 Pilot
Acronym: PAUSE2rctP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, James Douketis, Dr. James Douketis-Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAUSE-2-PILOT-2019
Record Dates: First submitted 2019-11-20; First posted 2019-12-10 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Atrial Fibrillation
Keywords: anticoagulant; atrial fibrillation; surgery; oral anticoagulant; high risk; blood thinner; DOAC; interruption; discontinue; elective; perioperative
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Patients taking apixaban, dabigatran, or rivaroxaban will be randomly assigned to follow 1) PAUSE or 2) ASRA perioperative DOAC management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Apixaban (Active Comparator): Patients currently taking apixaban that have atrial fibrillation and require an elective high-bleed-risk surgery/neuraxial anesthesia.
  Interventions: Other: PAUSE Perioperative DOAC Management; Other: ASRA Perioperative DOAC Management
- Dabigatran (Active Comparator): Patients currently taking dabigatran that have atrial fibrillation and require an elective high-bleed-risk surgery/neuraxial anesthesia.
  Interventions: Other: PAUSE Perioperative DOAC Management; Other: ASRA Perioperative DOAC Management
- Rivaroxaban (Active Comparator): Patients currently taking rivaroxaban that have atrial fibrillation and require an elective high-bleed-risk surgery/neuraxial anesthesia.
  Interventions: Other: PAUSE Perioperative DOAC Management; Other: ASRA Perioperative DOAC Management

INTERVENTIONS:
Other: PAUSE Perioperative DOAC Management — Apixaban & Rivaroxaban: Hold DOAC for 2 days before procedure. Re-start DOAC 2+ days post-procedure.
  Dabigatran (see below):
  CrCl ≥50: Hold DOAC for 2 days before procedure. Re-start DOAC 2+ days post-procedure.
  CrCl <50: Hold DOAC for 4 days before procedure. Re-start DOAC 2+ days post-procedure.
Other: ASRA Perioperative DOAC Management — Apixaban & Rivaroxaban: Hold DOAC for 3 days before procedure. Re-start DOAC 1+ days post-procedure.
  Dabigatran (see below):
  CrCl >80: Hold DOAC for 3 days before procedure. Re-start DOAC 1+ days post-procedure.
  CrCl 50-80: Hold DOAC for 4 days before procedure. Re-start DOAC 1+ days post-procedure.
  CrCl 30-49: Hold DOAC for 5 days before procedure. Re-start DOAC 1+ days post-procedure.
  *Low-dose heparin bridging can be used if at high A-TE risk

SUMMARY:
The proposed PAUSE-2 RCT study is the logical next step to the Perioperative Anticoagulant Use for Surgery Evaluation (PAUSE) study, which was completed on August 31, 2018. Both studies address the perioperative management of patients with atrial fibrillation (AF) who are receiving a direct oral anticoagulant (DOAC) and require an elective surgery/procedure. PAUSE did not address safe management of patients having a high-bleed-risk surgery/neuraxial anesthesia in whom there is concern about bleeding, especially neuraxial-related epidural hematomas that can lead to paralysis; such patients are often managed by the approach recommended by the American Society of Regional Anesthesia (ASRA). In PAUSE-2, investigators will test the hypothesis: (i) for patients having a high-bleed-risk surgery/neuraxial anesthesia, the simpler "PAUSE management" is as safe (non-inferior) to the more complex "ASRA management". PAUSE-2 will establish a standard for perioperative DOAC management in patients having high-bleed-risk surgery or neuraxial anesthesia.

To start, this will be a pilot study of a larger PAUSE-2-RCT. The investigators will be conducting this pilot study to assess the feasibility of the study at this smaller scale.

DETAILED DESCRIPTION:
The proposed PAUSE-2 RCT study is the logical next step to the Perioperative Anticoagulant Use for Surgery Evaluation (PAUSE) study, which was completed on August 31, 2018 and presented at the American Society of Hematology Conference on December 4, 2018. Both studies address the perioperative management of patients with atrial fibrillation (AF) who are receiving a direct oral anticoagulant (DOAC) (apixaban, dabigatran or rivaroxaban) and require an elective surgery/procedure. Standardized, DOAC-specific perioperative management is needed to: (i) minimize patient harm related to serious perioperative adverse events, comprising arterial thromboembolism (A-TE) and major bleeding (MB); and (ii) allow consistent, cost-efficient management that avoids cancelled surgeries/procedures and the need to reverse DOACs. PAUSE did not address safe management of patients having a high-bleed-risk surgery/neuraxial anesthesia in whom there is concern about bleeding, especially neuraxial-related epidural hematomas that can lead to paralysis; such patients are often managed by the approach recommended by the American Society of Regional Anesthesia (ASRA).

In PAUSE-2, the primary question is: (i) In patients having a high-bleed-risk surgery/neuraxial anesthesia, is the simple, shorter-DOAC-interruption PAUSE management as safe as the more complex, longer-interruption ASRA approach? Hypothesis: PAUSE management is non-inferior to ASRA management with expected perioperative risks in both groups of 2.5% for MB (2% non-inferiority margin) and 0.5% for A-TE (1% non-inferiority margin).

In PAUSE-2, the secondary question is: (i) are the PAUSE and ASRA management approaches associated with similar proportions of patients with minimal-to-no residual DOAC levels at surgery, and similar adherence to the DOAC interruption/resumption protocols? Exploratory postulate: PAUSE and ASRA approaches will have similar proportion of patients (±5%) with DOAC levels (<30, 30-49.9, and ≥50 ng/mL), and protocol adherence to perioperative DOACs interrupted and resumed.

Approximately 201 patients will be recruited for the PAUSE-2 Study pilot. This is 10% of the proposed main study (2,010 participants).

In all patients, a 5 mL blood sample will be taken just before surgery (but will be not available for clinical use and cannot be used for genetic testing). Plasma will be frozen and stored at each clinical site before shipment to the core laboratory at McMaster University for storage and standardized DOAC level measurement.

A focused patient enrolled before the procedure and followed up every week up to completion of their participation at 4 weeks (±5 days). Patients will be enrolled over a 1 year period.

To start, this will be a pilot study of a larger PAUSE-2-RCT. Conducting this pilot study will help assess the feasibility and methodology of the study at this smaller scale. It is important to evaluate the feasibility of recruitment, randomization and retention. As well, investigators need to assess the methodology and implementation of the randomized trial.

Note that the outcome for the pilot study is not to evaluate the safety of the perioperative procedure, but to examine the approach to be used in the intended larger study. The outcomes for the larger study will still be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥18 years) with AF/flutter who is receiving a DOAC: apixaban 2.5 mg or 5 mg BID; dabigatran 110 mg or 150 mg BID; or rivaroxaban 15 mg or 20 mg QD.
* Undergoing an elective surgery/procedure associated with a high-bleed-risk or any surgery/procedure requiring neuraxial anesthesia (includes regional blocks)
* Patient and their clinician are willing to adhere to DOAC interruption/continuation protocols.
* Patient to resume DOAC after surgery/procedure (i.e., no intent to discontinue DOAC).

Exclusion Criteria:

* Creatinine clearance (CrCl) <30 mL/min (dabigatran, rivaroxaban) and <25 mL/min (apixaban) based on the Cockroft-Gault equation, which is recommended for DOAC dosing.
* Patient taking a DOAC that is infrequently used (i.e., edoxaban, <5% Canadian DOAC market share in 2018) or is not available for clinical use in Canada or Europe (i.e., betrixaban).
* Patient taking a DOAC for a non-AF clinical indication (excluded to maintain study population homogeneity).
* Cognitive impairment or psychiatric illness that precludes collection of follow-up data.
* Inability or unwillingness to provide informed consent.
* Previous participation in PAUSE-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who had a major bleed | Each patient will be followed up every 7 days up to completion at 28 days post procedure date
  ≥1 of the criteria below:
  * bleeding that is fatal or is symptomatic and retroperitoneal, intracranial, intraspinal, intraocular, pericardial, intramuscular with compartment syndrome, or intra-articular
  * non-surgical bleeding causing a drop in hemoglobin ≥20 g/L (1.24 mmol/L) or leading to transfusion ≥2 units whole blood or red cells within 48 hours of the bleed
  * surgical bleed that leads to intervention (e.g., re-operation) or has one of: (i) interferes with mobilization; (ii) leads to delayed wound healing; or (iii) leads to deep wound infection
  * surgical site bleeding that is unexpected and prolonged and/or sufficiently large to cause hemodynamic instability associated with: (i) drop in hemoglobin ≥20 g/L (1.24 mmol/L); or (ii) transfusion of ≥2 units whole blood or red cells within 48 hours of the bleed
Number of patients who had an Arterial Thromboembolism (ATE) | Each patient will be followed up every 7 days up to completion at 28 days post procedure date
  Any of the following: stroke, systemic embolism, and/or transient ischemic attack.
  * Ischemic stroke: any new focal neurologic deficit that persists for >24 hours or any new focal neurologic deficit of any duration, that occurs with evidence of acute infarction on computed tomography (CT) or magnetic resonance imaging (MRI) of the brain.
  * Systemic embolism: symptomatic embolism to upper or lower extremity or abdominal organ, confirmed intra-operatively or by objective imaging (e.g., CT angiography).
  * Transient ischemic attack: symptomatic focal neurologic deficit (lasting typically <1 hour), that occurs with no evidence of acute infarction on CT/MRI of brain.

SECONDARY OUTCOMES:
Number of patients who died | Each patient will be followed up every 7 days up to completion at 28 days post procedure date
  Death due to any cause.
Number of patients who had a Clinically Relevant Non-Major Bleed | Each patient will be followed up every 7 days up to completion at 28 days post procedure date
  any overt bleeding not satisfying the criteria for major bleeding but considered clinically important with one or more of the following criteria met:
  * Requires minimal medical intervention (blood in urine or stool that is ongoing and requires a sigmoidoscopy, cystoscopy, CBI etc.) by a healthcare professional
  * Lead to hospitalization or increased level of care
  * Prompted a face-to-face (ie. not telephone, electronic) evaluation by a physician (this does not include visits prompted by pain, infection, other symptoms etc.)
Number of patients who had a Minor Bleed | Each patient will be followed up every 7 days up to completion at 28 days post procedure date
  Any overt bleeding not satisfying the criteria for major and clinically relevant non-major bleeding.
Number of patients who had a Venous Thromboembolism (VTE) | Each patient will be followed up every 7 days up to completion at 28 days post procedure date
  Any of the following: symptomatic deep vein thrombosis and/or pulmonary embolism, confirmed by objective imaging studies (e.g., ultrasound, CT pulmonary angiogram).
Number of patients who had an Acute Coronary Syndrome | Each patient will be followed up every 7 days up to completion at 28 days post procedure date
  Symptomatic myocardial ischemia, defined by pre-specified clinical and objective EKG- and/or troponin-related criteria.

OTHER OUTCOMES:
Concentrations of Anti-factor Xa | Pre-op day 0
  Measurement of pre-operative DOAC levels
Rate of Diluted Thrombin Time (dTT) | Pre-op day 0
  Measurement of pre-operative DOAC levels
Adherence to the DOAC interruption and resumption protocols | Approximately 1 week pre-op up to completion at 28 days post procedure date
  Measured by the number of days adhering to DOAC interruption and resumption protocols.

CONTACTS AND LOCATIONS:
Overall Officials: James D Douketis, MD, Principal Investigator — McMaster University/St. Joseph's Healthcare
Locations (3):
- Canada (3):
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario